CLINICAL TRIAL: NCT04119713
Title: Mechanisms of Immunotoxicology in Cancer Patients
Brief Title: Autoimmunity After Checkpoint Blockade
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 832823
Record Dates: First submitted 2019-09-23; First posted 2019-10-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Autoimmunity; Cancer; Immunotoxicity; Oncology
MeSH Terms: conditions — Autoimmune Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50 mls of peripheral blood will be drawn at the time that patients are prescribed an immune checkpoint inhibitor (ICI) which will be banked for serum and PBMCs. No more than 50 mls of blood will be drawn at the following established points: at the time of the second drug infusion, at 6 months, at 12 months, and between 18 and 24 months. Additionally, no more than 50 mls of blood will be drawn at any time that a participant develops an autoimmune complication.
  An assessment tool that queries symptoms suggestive of a number of common immunotherapy-related adverse events (PRO-CTCAE) will be administered to consented patients at each visit in concert with the standard-of-care patient reported outcomes tool currently in use in Cancer Center clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Adult patients with a diagnosis of cancer receiving checkpoint inhibitor therapy at the University of Pennsylvania's Abramson Cancer Center (ACC).

SUMMARY:
The purpose of this study is to better understand how the treatment of cancer with immune checkpoint inhibitors (ICI) leads to the development of autoimmunity. Specifically, we wish to understand the genetics and immune system features that cause a subset of cancer patients treated with checkpoint inhibitor therapy to develop an immune-related adverse event (irAE).

DETAILED DESCRIPTION:
The goal of this study is to understand how the treatment of cancer with checkpoint inhibitors leads to the development of autoimmunity. Specifically, to understand the genetics and immune system features that cause a subset of cancer patients treated with checkpoint inhibitors to develop autoimmunity. At least 300 patients will be enrolled when they are initially prescribed any checkpoint inhibitor. Peripheral blood and serum from patients when they enroll and examine the genetics, serum factors, and phenotype of the immune system. There is no planned intervention. Subjects will be asked to provide peripheral blood and serum at established time points when they are getting therapeutic infusions and routine clinical labs, as well as, at the time they develop any autoimmune symptoms. Urine may also be collected at the time of enrollment, standard study visits, and/or at the time of an autoimmune complication. Inclusion criteria include a diagnosis of cancer, prescription for a checkpoint inhibitor, and fluency in English. Exclusion criteria include any subjects not willing or able to give consent, children under the age of 18, and history of transplant. There will not be any interventions. Clinical data will be extracted from electronic medical records. Coded data will be stored in a REDCap database. Protected health information (PHI) and study key stored at UPenn on a password-protected database on an encrypted drive that is institutionally secured and managed by the University of Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer and prescription for a checkpoint inhibitor

Exclusion Criteria:

* Any subjects not willing or able to give consent
* Children under the age of 18
* A history of transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are able to consent to the study and are identified by their physician or a clinical coordinator to receive an immune checkpoint inhibitor for the treatment of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The phenotype and function of peripheral blood cells (i.e., CD4+ T cells, CD8+ T cells, B cells, myeloid cells) characteristic to patients receiving checkpoint inhibitor therapy. | 6 years
  The phenotypic analysis will include multiple surface markers that define populations of cells, including activated, memory, and regulatory populations. Cells will also be activated to determine which cytokines are produced.
The prevalence of immune-related adverse events (irAEs) that complicate checkpoint inhibitor therapy. | 6 years
  This is a pilot analysis to better understand how the treatment of cancer with immune checkpoint inhibitors leads to the development of autoimmunity in a subset of cancer patients.

SECONDARY OUTCOMES:
The number of future research studies and/or collaborations resulting directly from the databank of tissues and other relevant clinical information that will be established. | 6 years
  To facilitate collaborations between research groups from diverse disciplines that enables rapid translation of ongoing and future basic research findings that leads to individualized, or personalized care for patients receiving immunotherapies.

CONTACTS AND LOCATIONS:
Overall Officials: Sokratis Apostolidis, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided